CLINICAL TRIAL: NCT02564757
Title: Does Pregnancy Increase Risk of Ventral Hernia Recurrence?
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Erling Oma, Research scholar, Bispebjerg Hospital
Other Study IDs: eoma2
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Recurrent Hernia of Anterior Abdominal Wall
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will examine if pregnancy increases risk of ventral hernia recurrence

DETAILED DESCRIPTION:
The investigators will establish a cohort of female fertile patients who underwent ventral hernia repair (Umbilical, Epigastric and Incisional hernia repair) registered in the Danish Hernia Database. The investigators will link these data at an individual level with the Danish National Patient Registry (DNPR), Danish Medical Birth Registry (DMBR) and the Danish Civil Registry (CPR).

From DMBR, subsequent pregnancies in the study cohort will be noted. From DNPR, ventral hernia recurrence, defined as clinical recurrence and/or reoperation for recurrence will be noted. Cases registered with both clinical recurrence and reoperation for recurrence, the date of the earliest registration will be defined as the date of ventral hernia recurrence.

From CPR, date of death or emigration will be noted.

Through an extended Cox regression analysis, handling pregnancy as a time-dependent variable, the investigators will examine whether pregnancy is associated with an increased risk of ventral hernia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Fertile female patient

Exclusion Criteria:

* non-Danish citizen

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fertile female patients who have undergone ventral hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 3578 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clinical Ventral Hernia (Epigastric, Umbilical and Incisional Hernia) Recurrence | 0-7 years
  Clinical ventral hernia recurrence will be defined as clinical recurrence retrieved from the Danish National Patient Registry.
Ventral Hernia (Epigastric, Umbilical and Incisional Hernia) Recurrence Repair | 0-8 years
  Ventral hernia recurrence repair will be defined as reoperation retrieved from the Danish National Patient Registry.

CONTACTS AND LOCATIONS:
Overall Officials: Lars N Jorgensen, MD, DMSc, Study Chair — Bispebjerg Hospital, University of Copenhagen